CLINICAL TRIAL: NCT03598686
Title: Home-based Plus Self-testing to Improve HIV Testing Coverage in Rural Lesotho - a Cluster Randomized Controlled Trial in Rural Lesotho.
Brief Title: HOme-based SElf-testiNG - a Cluster Randomized Controlled Trial in Rural Lesotho (HOSENG)
Acronym: HOSENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tracy Glass (Other)
Collaborators: SolidarMed (Other); Ministry of Health, Lesotho (Other Government); University of Basel (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Tracy Glass, Head of Statistics, Principal Investigator, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P002-18-3.0
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: HIV; HIV/AIDS
Keywords: HIV; HIV/AIDS; self-testing; HIVST; home-based; community-based; lesotho; oraquick; testing coverage; htc campaign
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The HOSENG study is linked to a follow-up trial, the VIBRA study. Together they are called the GET ON ("GETing tOwards Ninety") research project. The HOSENG study with its home-based HIV testing campaign provides the platform for the VIBRA study. The reasons for this interlinked design are: a) potential study participants for VIBRA trial (HIV-positive individuals not on ART) are recruited during the HOSENG study, b) this design allows us to assess the entire HIV/AIDS care cascade in one larger project, and c) both trials rely on interventions involving VHWs, who need to be randomized and specifically trained. Therefore, it is more efficient and feasible to run both trials parallel and randomize at one time point.
  The HOSENG study is a cluster randomized, parallel-group (1:1:1:1 allocation), open-label, superiority, prospective clinical trial. Clusters are stratified by district, size of village, and village access to the nearest health facility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOSENG Control (No Intervention): Standard of care during a door-to-door HIV testing campaign:
  1. For present household members: blood-based HIV testing
  2. For absent household members or household members who refuse testing: They are encouraged to get tested by the Village Health Worker (VHW) or the nearby health facility
- HOSENG Intervention (Experimental): HOSENG Intervention during a door-to-door HIV testing campaign:
  1. For present household members: blood-based HIV testing
     a) If any absent person in the household: One of the present household members is tested and trained using the oral HIVST (OraQuick©)
  2. For absent household members or household members who refuse testing: One oral HIVST (OraQuick©) is left behind and has to be brought back to the VHW after usage. Otherwise it will be collected by the VHW after two weeks.
  Interventions: Diagnostic Test: OraQuick

INTERVENTIONS:
Diagnostic Test: OraQuick — Most trials assessing oral HIVST make use of OraQuick® (OraQuick ADVANCE HIV I/II test kits, packaged for self-use), an oral-fluid rapid self-test. OraQuick® is a 2nd generation serology assay with a sensitivity of 99.3% (95%CI; 98.4%, 99.7%) and a specificity of 99.8% (95%CI; 99.6%, 99.9%). In a pilot study with 59 participants conducted in Lesotho in 2015 more than 90% of the participants found utilization of OraQuick® easy, and trusted the results of the self-test kit. The WHO recently has announced that OraQuick becomes the first prequalified HIV self-test, in order to improve diagnosis in low-resourced health systems and in countries where stigma prevents people from getting tested. Therefore, OraQuick® is now available in Lesotho for as little as 2 USD per test kit.
  Arms: HOSENG Intervention

SUMMARY:
This cluster-randomized trial aims to evaluate the efficacy of the use of oral HIV self-testing (HIVST) among individuals who are absent or who decline HIV testing during home-based HIV testing

DETAILED DESCRIPTION:
By launching the 90-90-90 strategy UNAIDS has shown a way forward in controlling and finally eradicating the deadly AIDS epidemic. Recent global data shows that progress towards the first UNAIDS target, i.e. to ensure that 90% of HIV-positive individuals are aware of their status, is lower than progress in other areas of the HIV care cascade. It is estimated that still approximately 2.7 million HIV-positive people do not know their HIV status.

Home- or community-based HIV testing has been proven to be very effective in resource-limited settings and therefore is a key strategy endorsed by WHO. Although acceptance of testing during such campaigns is usually very high, coverage remains low due to absent household members. And usually these absent people are men and young adults - both of which have a disproportionately high risk of HIV acquisition and poorer clinical outcomes once infected.

Oral HIV self-testing (HIVST) has shown to be an accurate diagnostic tool with a high acceptance and feasibility in sub-Saharan Africa. Experiences from the sub-Saharan region suggest that when HIV self-testing is provided as part of a home-based HIV testing campaigns, it can increase uptake of testing and facilitate linkage to care, especially among individuals who are at high risk of HIV infection.

The HOSENG study is linked to a follow-up trial, the VIBRA study. Together they are called the GET ON ("GETing tOwards Ninety") research project. The HOSENG study with its home-based HIV testing campaign provides the platform for the VIBRA study.

The HOSENG study is a cluster randomized, parallel-group (1:1:1:1 allocation), open-label, superiority, prospective clinical trial. Clusters are stratified by district, size of village, and village access to the nearest health facility.

The primary endpoint is HIV testing coverage among individuals aged 12 years or older in the surveyed area within 120 days after the home visit, defined as the proportion of all individuals 12 years or older living in a household of the surveyed area with a confirmed HIV test result. The secondary enpoints are listed below.

For the entire GET ON project we will collect cost data. Specifically for HOSENG trial, first, direct costs of the intervention will be assessed: Staff costs (campaign team, VHWs, clinic staff), personnel training costs (VHWs), cost of equipment (HIV tests, consumables, logistics), as well as non-medical costs to the participant (i.e. cost of transportation to ART service). These data will provide the average cost per participant achieving the primary endpoint within 120 days in each cluster arm ('per participant tested cost'). Secondly, a cost-effectiveness analysis will be performed with respect to the primary endpoint. Da-ta to assess patient level costs will be collected from a randomly selected sub-sample of study participants from each cluster arm. Costs will be reported as means (incl. SD) and medians (incl. IQRs) in local currencies and US dollars and International Dollars.

A nested study (ADORE study: "ADolescent ORal sElf-testing") will explore the acceptability of oral HIVST among adolescents and young adults with quantitative methods (see secondary endpoint) and qualitative methods: A qualitative case-control study. Cases are those who refused testing through oral HIVST and controls are those who accepted testing through oral HIVST. We plan to conduct at least 10 interviews per group, stratified by two pre-defined factors (male vs female; age 12-15 vs age 16-24), following the concept of saturation. Data will be collected by a trained study member, who was part of the HIV testing campaign, using a piloted interview questionnaire (KoboToolbox; www.kobotoolbox.org), conducted in the local language (Sesotho). Qualitative data will be recorded, transcribed, translated into English and coded and analyzed using the Framework Method.

More, detailed information:

* https://getonproject.wordpress.com
* https://www.swisstph.ch/en/topics/hiv-aids/

ELIGIBILITY:
Eligibility - clusters

Inclusion criteria:

1. the cluster is rural and clearly confined to the catchment area of one of the study clinics i. one cluster usually consists of one village, but could include several small villages serviced by the same VHW
2. the cluster has at least one registered VHW who is willing to participate and fulfills the following criteria: i. is at least 18 years of age ii. has adequate reading and writing skills iii. successfully passes the training assessment, assessed by a local person independent to GET ON research project and GET ON research team. Two criteria have to be fulfilled: a. is able to fill in the assessment (tick boxes, write in correct fields) b. is able to give an adequate answer regarding open question (in order to see if VHW is able to read and write and has a basic logic thinking)

Exclusion criteria:

1. village authority (=village chief) opposed to trial participation (verbal assent)
2. VHW opposed to trial participation or not fulfilling the minimum requirements mentioned above (=inclusion criteria, point b) i. Note: if a cluster entails several VHWs, then the cluster can still participate if there is at least one VHW in the cluster who is willing to trial participation and fulfills the minimum requirements.

Eligibility - household

Inclusion criteria:

a) signed informed consent form from household head or representative aged 18 years or older

Exclusion criteria:

a) no signed informed consent form from household head or representative

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
HIV testing coverage | within 120 days after enrolment (i.e. HTS campaign)
  HIV testing coverage among individuals aged 12 years or older in the surveyed area within 120 days after the HIV testing and service (HTS) campaign, defined as the proportion of all individuals 12 years or older living in a household of the surveyed area with a confirmed HIV test result

SECONDARY OUTCOMES:
HIV testing coverage among adolescents and young adults (ADORE nested study outcome) | within 120 days after enrolment (i.e. HTS campaign)
  HIV testing coverage among 12-24 years old individuals in the surveyed area within 120 days after the HTS campaign, defined as the proportion of all 15-24 years old individuals living in a household of the surveyed area with a confirmed HIV test result.
Blood-based HIV testing uptake | at enrolment (i.e. HTS campaign)
  Blood-based HIV testing uptake, defined as the proportion of all individuals living in a household of the surveyed area, being eligible for blood-based HIV testing and accepting to be tested using blood-based point-of-care HIV test during the home-visit.
Oral HIVST uptake using OraQuick | at enrolment (i.e. HTS campaign) and within 120 days after enrolment (i.e. HTS campaign)
  Oral HIVST uptake among absent individuals, defined as the proportion of all individuals living in a household of the surveyed area for whom an oral HIVST was left behind and who accepted to be self-tested using the oral HIVST.
Overall HIV testing coverage | within 120 days after enrolment (i.e. HTS campaign)
  HIV testing coverage irrespective of age, defined as the proportion of all individuals living in a household of the surveyed area with a confirmed HIV test result

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, MD, Study Director — Swiss TPH; Manuel Battegay, MD, Study Chair — University Hospital, Basel, Switzerland; Josephine Muhairwe, MD, Study Chair — SolidarMed; Tracy R Glass, PhD, Principal Investigator — Swiss TPH
Locations (2):
- Lesotho (2):
  - District of Butha-Buthe, Butha-Buthe
  - District of Mokhotlong, Mokhotlong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amstutz A, Matsela L, Lejone TI, Kopo M, Glass TR, Labhardt ND. Reaching Absent and Refusing Individuals During Home-Based HIV Testing Through Self-Testing-at What Cost? Front Med (Lausanne). 2021 Jun 29;8:653677. doi: 10.3389/fmed.2021.653677. eCollection 2021. PMID 34268321
- [Derived] Amstutz A, Lejone TI, Khesa L, Muhairwe J, Bresser M, Vanobberghen F, Kopo M, Kao M, Nsakala BL, Tlali K, Klimkait T, Battegay M, Labhardt ND, Glass TR. Home-based oral self-testing for absent and declining individuals during a door-to-door HIV testing campaign in rural Lesotho (HOSENG): a cluster-randomised trial. Lancet HIV. 2020 Nov;7(11):e752-e761. doi: 10.1016/S2352-3018(20)30233-2. Epub 2020 Oct 9. PMID 33045193
- [Derived] Amstutz A, Kopo M, Lejone TI, Khesa L, Kao M, Muhairwe J, Glass TR, Labhardt ND. "If it is left, it becomes easy for me to get tested": Use of oral self-tests and community health workers to maximize the potential of home-based HIV testing among adolescents in Lesotho. J Int AIDS Soc. 2020 Sep;23 Suppl 5(Suppl 5):e25563. doi: 10.1002/jia2.25563. PMID 32869527
- [Derived] Amstutz A, Lejone TI, Khesa L, Muhairwe J, Nsakala BL, Tlali K, Bresser M, Vanobberghen F, Kopo M, Kao M, Klimkait T, Battegay M, Labhardt ND, Glass TR. The HOSENG trial - Effect of the provision of oral self-testing for absent and refusing individuals during a door-to-door HIV-testing campaign on testing coverage: protocol of a cluster-randomized clinical trial in rural Lesotho. Trials. 2019 Aug 13;20(1):496. doi: 10.1186/s13063-019-3469-2. PMID 31409421
- See also: Official Project Homepage — http://getonproject.wordpress.com/